CLINICAL TRIAL: NCT05096455
Title: Hypertriglyceridemia Associated Acute Pancreatitis in Intensive Care Unit and Therapeutic Plasmapheresis: a Multicenter Retrospective Study
Brief Title: Hypertriglyceridemia Associated Acute Pancreatitis in Intensive Care Unit and Therapeutic Plasmapheresis
Acronym: TRIPAN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2021/SB-01
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Pancreatitis; Hypertriglyceridemia
Keywords: ICU
MeSH Terms: conditions — Pancreatitis; Hypertriglyceridemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- severe acute pancreatitis: Patients 18 years of age or older admitted to intensive care or resuscitation for severe acute pancreatitis (AP) with hypertriglyceridemia (HTG)

SUMMARY:
Acute pancreatitis (AP) is a one of the potentially life-threatening complication of severe hypertriglyceridemia (HTG), with mortality around to 30%.

HTG-associated PA and their complications management has to be the same as the other pancreatitis, but they are associated with the worse clinical outcomes. Triglycerides levels are correlated with the risk of pancreatitis and severity.

Therapeutic plasma exchange (TPE) could provide positive effects in reducing triglyceridemia plasma levels during the acute phase of HTG-AP, and in prevention of recurrence. There is currently no difference about mortality in studies. Some authors have recommended its use only in severe HTG-AP and have precised the need of early initiation to have positive results.

Despite such promising findings from studies, the effects of therapeutic plasma exchange on HTG-associated PA have never been specifically assessed and its benefits in critically ill patients with AP remains uncertain.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Admission in ICU for acute pancreatitis associated with HTG

Exclusion Criteria : Patient without norepinephrine or missing data.

* Acute pancreatitis without HTG
* Patient already include in this study
* Patient opposed to use of his data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient hospitalized with severe acute pancreatitis of hypertriglycemic origin admitted to the ICU between January 2010 and January 2020.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality at Day 28 | Day 28
  Assess the factors on admission associated with the prognosis of patients admitted in ICU for HTG-associated PA.
  Factors associated with death at D28 will be considered individually for entry into a multivariate model. The following variables of interest will be tested in the model: SOFA score, triglyceride level at admission, obesity.

SECONDARY OUTCOMES:
Length of hospitalization | Day 28
  Describe length of stay in ICU and on hospital for patients admitted in ICU for HTG-associated PA
Use of organ support | Day 28
  Describe use of organ supports (vasopressors, extra-renal dialysis and mechanical ventilation)
Assess benefit of plasmapheresis | Day 28
  Assess benefit of plasmapheresis for patients admitted in ICU for HTG-associated PA

CONTACTS AND LOCATIONS:
Overall Officials: stephanie Bulyez, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France